CLINICAL TRIAL: NCT06771414
Title: Metagenomic Characterization of the Intestinal Microbiota in ALS Patients and Association With Clinical Phenotypes
Acronym: ALS-Gut
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); ARSLA (Unknown); ALS Association (Other); Filière FilSLAN (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP241702
Record Dates: First submitted 2024-12-20; First posted 2025-01-13 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2024-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Amyotrophic Lateral Sclerosis; microbiota; gut microbiota; french gut
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: data collection — data collection

SUMMARY:
"Amyotrophic lateral sclerosis (ALS) is a progressive neurodegenerative disease involving motor neurons in the cerebral cortex, brain stem and spinal cord. Loss of functional motor neurons is responsible for rapid progressive muscle paralysis, generally leading to death from respiratory failure within 3 to 5 years. Data obtained in mouse models of the disease suggest that changes in the intestinal microbiota may be involved in the pathophysiology of the disease. However, to date, there are no solid data on the existence of intestinal dysbiosis in ALS patients and its prognostic influence. The ALS-Gut study will make it possible for the first time to quantitatively and qualitatively characterize the gut microbiota in a large population of French ALS patients, and to identify changes associated with the disease compared with healthy subjects. It will also identify possible associations between observed deviations in microbiota and the ALS phenotype, its management modalities, and its evolutionary profile. This study will thus pave the way for innovative therapeutic strategies aimed at re-establishing a favorable gut microbiota profile, in order to limit the progression of motor impairment.

The aim of the ALS-Gut study is to quantitatively and qualitatively characterize the microbiota in a cohort of 300 French ALS patients, and to correlate these results with the clinical features of the disease. The ALS-Gut study will be based on the "Le French Gut" project carried out by a consortium comprising INRAE, AP-HP, INSERM and Institut Pasteur on 100,000 volunteers, aimed at characterizing the heterogeneity and diversity of the intestinal microbiota of subjects living in France.

The ALS-Gut study is a non-human research study, which will use clinical data collected prospectively in 18 French ALS expert centers as part of the routine management of 300 French ALS patients participating in the "Le French Gut" project."

DETAILED DESCRIPTION:
"The ALS-Gut study aims to quantitatively and qualitatively characterize the microbiota in a cohort of 300 French ALS patients, and to correlate these results with the clinical features of the disease.

The ALS-Gut study will build on the "Le French Gut" project conducted by a consortium comprising INRAE, AP-HP, INSERM and Institut Pasteur on 100,000 volunteers, aimed at characterizing the heterogeneity and diversity of the gut microbiota of subjects living in France (https://lefrenchgut.fr). The "French Gut" is a non-interventional study (protocol appended) involving human subjects. It is prospective, nationwide, with the creation of a biological collection (faeces) linked to the exploitation of data from questionnaires and the ""Système National des Données de Santé"" (SNDS). Following volunteer registration via the study's dedicated website, a stool sample will be taken at home for analysis of the fecal microbiota by shotgun metagenomic sequencing. The various components of the microbiota will then be compared with individual data obtained from specific questionnaires, completed on the French Gut website by the volunteer, such as dietary habits or current state of health.

The ""French Gut"" project will map the healthy gut microbiota in France, and also describe variations in gut microbiota associated with the presence and development of certain diseases, particularly neurodegenerative diseases such as ALS.

The ALS-Gut study is a non-human research study, which will use clinical data collected prospectively in 18 French ALS expert centers as part of the routine management of 300 French ALS patients participating in the "Le French Gut" project.

The clinical data collected as part of the ALS-Gut study will be analyzed in conjunction with the metagenomic results obtained by INRAE, based on a stool sample sent to the French Gut consortium by the patient in advance, on a voluntary basis."

ELIGIBILITY:
Common inclusion criteria :

1. Patient with ALS that is possible, probable with the support of complementary examinations, clinically probable or defined according to the revised El Escorial diagnostic criteria (Brooks, et al. 2000).
2. Follow-up in one of the 18 French ALS expert centers participating in the study.
3. Age ≥18 years
4. Social security affiliation or beneficiary
5. Informed of the ALS-Gut study and not objecting to the collection of his/her data

Common non-inclusion criteria:

1. Other concomitant neurodegenerative pathology
2. Persons subject to a protective measure, notably guardianship or trusteeship, or unable to express their consent.

PATIENTS ALREADY INCLUDED IN FRENCH GUT 1. Patient agrees to provide French Gut with his or her participation number.

PATIENTS NOT YET INCLUDED IN FRENCH GUT

Inclusion criteria specific to patients not included in the French Gut study :

1. Patient agreeing to take part in the French Gut project, i.e. registering on his or her own initiative, on the project's dedicated website (https://lefrenchgut.fr/) and completing a detailed questionnaire. Then, on receipt of the stool sampling kit at home, return the stool sample to INRAE.

Specific non-inclusion criteria for patients not included in the French Gut (criteria linked to the French Gut) :

1. Person not living in France
2. Person who has had a colectomy (declarative) ;
3. Person with a digestive stoma (declarative);
4. Colonoscopy performed in the 3 months prior to inclusion (declarative).
5. Antibiotics taken in the 3 months prior to inclusion (self-reported);

Secondary exclusion criteria specific to patients included in the ALS-Gut study prior to inclusion in French Gut

1. No response to the French Gut entry questionnaire
2. Failure to send a compliant stool sample
3. Person who has not signed a French Gut consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ALS
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
characterize the intestinal microbiota of French ALS patients | Day 0
  description of the presence and abundance in the samples of each of the 10.4 million gut microbial genes listed in the IGC2 (Integrated Gene Catalog 2) catalog

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.